CLINICAL TRIAL: NCT07189078
Title: IntHyx : Intubation Strategies for Patients With Acute Hypoxemic Respiratory Failure
Acronym: IntHyx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49RC24_0293; 2025-A01380-49 (Other: French National Drug Regulatory Authority (ANSM))
Record Dates: First submitted 2025-08-29; First posted 2025-09-23 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: Randomization; Intubation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Liberal" intubation strategy (Experimental): Endotracheal intubation is recommended if SpO₂/FiO₂ < 110 for more than 5 minutes.
  In addition, intubation is also recommended in the liberal strategy if any of the restrictive strategy criteria occur and persist for more than 5 minutes.
  Interventions: Procedure: Liberal intubation strategy
- Restrictive intubation strategy (Experimental): Endotracheal intubation is recommended only if at least one of the following criteria persists for more than 5 minutes:
  1. Respiratory rate > 40/min, persistent use of accessory muscles, or thoracoabdominal paradox.
  2. SpO₂/FiO₂ < 88.
  3. Neurological or systemic impairment attributable to hypoxemia, defined as: altered higher brain functions without another identifiable cause, Glasgow Coma Scale ≤ 12, uncontrolled hemodynamic instability, or rising lactate levels.
  Interventions: Procedure: Restrictive intubation strategy

INTERVENTIONS:
Procedure: Restrictive intubation strategy — Endotracheal intubation is recommended only if at least one of the following criteria persists for more than 5 minutes:
  1. Respiratory rate > 40/min, persistent use of accessory muscles, or thoracoabdominal paradox.
  2. SpO₂/FiO₂ < 88.
  3. Neurological or systemic impairment attributable to hypoxemia, defined as: altered higher brain functions without another identifiable cause, Glasgow Coma Scale ≤ 12, uncontrolled hemodynamic instability, or rising lactate levels.
  Arms: Restrictive intubation strategy
Procedure: Liberal intubation strategy — Endotracheal intubation is recommended if SpO₂/FiO₂ < 110 for more than 5 minutes.
  In addition, intubation is also recommended in the liberal strategy if any of the restrictive strategy criteria occur and persist for more than 5 minutes.
  Arms: "Liberal" intubation strategy

SUMMARY:
Acute hypoxemic respiratory failure requires endotracheal intubation and invasive mechanical ventilation in approximately 30-40% of cases, due to severe hypoxemia and/or clinical signs of acute respiratory distress. The primary objectives of invasive mechanical ventilation are to reduce respiratory effort and improve oxygenation. However, this intervention is also associated with both direct and indirect adverse effects, mainly linked to the need for sedation and often neuromuscular blockade. These include hemodynamic compromise, neuromuscular weakness, ventilator-induced lung injury, and infectious complications.

An ideal intubation strategy would therefore strike a balance: avoiding the risks of delayed intubation-such as refractory hypoxemia, excessive respiratory effort, and patient self-inflicted lung injury (P-SILI)-while limiting complications associated with invasive mechanical ventilation by withholding it in patients who might otherwise recover without. To date, the optimal strategy for achieving this risk-benefit balance remains uncertain.

Clinical practice suggests a broad consensus on the necessity of intubation when so-called safety criteria are met: severe hypoxemia (SaO₂/FiO₂ ratio < 88), marked respiratory distress (use of accessory muscles, thoracoabdominal paradox, respiratory rate > 40/min), extra-respiratory manifestations of hypoxia (e.g., altered consciousness), and/or uncontrolled hemodynamic instability. Beyond these safety thresholds, however, debate persists. Some advocate for earlier intubation-a so-called liberal approach-triggered by predefined hypoxemia criteria (e.g., SpO₂/FiO₂ < 110), with the aim of limiting the deleterious consequences of sustained hypoxemia.

In routine practice, the criteria guiding intubation vary widely between clinicians and cannot be attributed to strong scientific evidence. This study therefore seeks to compare, in a randomized interventional design, the two main strategies currently applied across centers:

* Liberal intubation strategy: prioritizing the prevention of organ dysfunction related to hypoxemia (notably hypoxic cardiac arrest) and the risk of P-SILI.
* Restrictive intubation strategy: prioritizing the reduction of invasive mechanical ventilation use, with the goal of minimizing ventilation-related harm and its associated therapeutic burden.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient admitted to intensive care less than 24 hours ago
* Acute respiratory failure with hypoxemia defined by either:

  * Oxygen therapy ≥ 10 L/min via high-concentration mask required for SpO2 ≥ 92%
  * High-flow oxygen therapy with FiO2 ≥ 50% required for SpO2 ≥ 92%
* Informed consent of the patient or a trusted relative (when the patient is unable to give consent)

Exclusion Criteria:

* Acute hypercapnic respiratory failure (defined by PaCO2 > 45 mmHg)
* Cardiogenic pulmonary edema
* Exacerbation of chronic respiratory disease
* Respiratory failure requiring long-term oxygen therapy
* Neuromuscular disease
* Glasgow Coma Scale score ≤ 12
* Decision to intubate immediately
* Invasive mechanical ventilation within the previous 7 days
* Treatment limitation decisions for intubation
* Person deprived of liberty by judicial or administrative decision : Person undergoing compulsory psychiatric care, person subject to legal protection measures, Pregnant, breastfeeding, or parturient patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Impact of a liberal intubation strategy compared to a restrictive strategy in regards to organ support duration, taking mortality into account | Day 28
  Composite endpoint consisting of death and number of days with organ failure at D28, analyzed using the Win Ratio method.

SECONDARY OUTCOMES:
Evaluate the impact of the intubation strategy on intubation rates over time. | Day 28
  Time of intubation (if performed).
Assess the impact of the intubation strategy on each component of the composite primary endpoint. | Day 28
  Components of the composite primary endpoint:
  * All-cause mortality
  * Duration of mechanical ventilation
  * Duration of vasopressor support
  * Duration of renal replacement therapy
Assess the impact of the intubation strategy on the severity of vital organ failure and the duration of care. | Day 28
  Measurements of SOFA score (points), Length of stay in the intensive care unit (days) and total hospital length of stay (days) SOFA is Sepsis-related Organ Failure Assessment : score range form 0 to 24, the higher scores indicating the the more severe condition
Assess the impact of the intubation strategy on quality of life at day 90. | Day 90
  5Level-EuroQuol-5Dimensions score (EQ-5D-5L). The scale measures quality of life on a 5-component scale. A health state of 11,111 indicate no problem in any dimension, a health state of 55,555 indicates extreme problems in every dimension
Assess the impact of the intubation strategy on the rate of procedure-related adverse events. | within 30 minutes of the start of the intubation procedure
  Endpoint: Occurrence, within 30 minutes of the start of the intubation procedure, of any of the following events:
  * SpO₂ decrease to less than 80%;
  * Hemodynamic instability (defined as: Systolic blood pressure <65 mmHg recorded at least once, or Systolic blood pressure <90 mmHg for more than 30 minutes despite adequate volume resuscitation, or New requirement for vasopressors or an increase in vasopressor dose by more than 30%)
  * Cardiac arrest;
  * Severe arrhythmia.
Assess the impact of the intubation strategy on the rate of adverse events related to invasive mechanical ventilation. | Day 28
  Occurrence, at any time up to day 28, of any of the following events:
  * Ventilator-associated pneumonia;
  * Pneumothorax;
  * Delirium (as assessed by CAM-ICU score).
Assess the impact of the intubation strategy on the rate of adverse events potentially related to delayed intubation. | Day 28
  Occurrence of any of the following events:
  * Cardiac arrest in a non-intubated patient;
  * Need for emergency intubation that could not be safely delayed by 10 minutes;
  * Aspiration pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde TAILLANTOU-CANDAU, Doctor, Principal Investigator — University Hospital, Angers
Locations (9):
- France (9):
  - Angers University Hospital, ICU, Angers
  - Le Mans Hospital, ICU, Le Mans
  - Nantes University Hospital, ICU, Nantes
  - Orléans University hospital, ICU, Orléans
  - Pitié-Salpétrière Hospital, Paris University Hospital, ICU, Paris
  - Guadeloupe University Hospital, ICU, Pointe à Pitre
  - Rennes University Hospital, ICU, Rennes
  - Tours University Hospital, ICU, Tours
  - Vannes Hospital, ICU, Vannes

IPD SHARING:
Plan to Share IPD: No